CLINICAL TRIAL: NCT05433493
Title: Effect of Individual Cognitive Stimulation on Memory and Executive Functioning in Older Adults With Mild to Moderate Alzheimer's Disease: A Multicentre Randomised Controlled Trial
Brief Title: Effect of Individual Cognitive Stimulation on Memory and Executive Function in Older Adults With Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rsocialform - Geriatria, Lda (Other)
Collaborators: Aveiro University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20220621
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2022-07

CONDITIONS: Dementia; Neurocognitive Disorders; Cognitive Impairment; Cognitive Dysfunction; Cognitive Decline
Keywords: older adults; cognitive function; memory; executive function; dementia; cognitive stimulation therapy; cognition; neurocognitive disorders; individual therapy; non-pharmacological therapy; randomised controlled trial; Alzheimer disease
MeSH Terms: conditions — Dementia; Neurocognitive Disorders; Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants who meet the inclusion criteria will be randomly assigned to the intervention group receiving individual CS or to the control group receiving treatment as usual (participating in the activities previously established in their individual intervention plan).
  Participants in the intervention group will participate in two individual CS sessions per week for 12 weeks in addition to their treatment as usual. The sessions will include the same protocol in every participant site.
  Interventions: Behavioral: Cognitive stimulation
- Control group (No Intervention): Participants in the control group will receive treatment/activities as usual, participating in the activities previously established in their individual intervention plan.

INTERVENTIONS:
Behavioral: Cognitive stimulation — The intervention program will have 24 sessions (base scheme of 4 series of 6 sessions), lasting approximately 45 min and will be developed according to the following structure: - welcoming (greeting to the participant) (5 min); - orientation to reality (10 min); - main cognitive stimulation activity (25 min); - return to calm and evaluation of the session (5 min).
  The CS sessions will have an individual format and will be conducted by a professional with experience in CS and previously trained in this intervention. The intervention sessions will include several activities based on the CS principles, with evidence suggesting positive participant effects. The CS sessions will be carried out using material, developed by the principal investigator, in digital format (power point presentations). There will be no repetition of activities, and throughout the base CS program, the degree of difficulty of the exercises will be adjusted based on the dementia stage of the participant.
  Arms: Intervention group

SUMMARY:
This multicentre study, with a randomised controlled repeated measures experimental design, will be conducted in several Portuguese institutions, which provide care and supportive services for older adults diagnosed with mild or moderate Alzheimer's disease (AD), with an aim to assess the effect of individual cognitive stimulation (CS) on memory and executive functioning. Participants in the intervention group will attend 24 individual CS sessions, twice weekly for 12 weeks. Participants in the control group will complete their usual routines without any activity restrictions.

DETAILED DESCRIPTION:
Neurocognitive disorders (NCD) currently affect around 55 million people worldwide and expected to increase to 78 million by 2030 and 139 million by 2050, with Alzheimer's disease (AD) potentially accounting for 60-70% of dementia cases. Dementia is a syndrome, generally chronic or progressive in nature, that causes deterioration of cognitive function, particularly memory and executive functions, beyond what is expected in normal aging. However, there is evidence that in the early stages of NCD, people can learn and improve their cognitive functions through interventions such as CS. CS is a psychosocial intervention and a non-pharmacological therapy recommended by international practice guidelines for people with mild-to-moderate stage AD. However, it is also important to investigate whether NCD generates new skills or only preserves acquired skills, given that AD manifests initially and notably with deficits in memory and learning, sometimes accompanied by deficits in executive functions. Testing the effectiveness of CS by recruiting a representative sample from several Portuguese districts and using a CS programme with detailed and comprehendible content, may elicit relevant evidence in clinical practice, contribute to the development of social development programs and initiatives to ensure social protection and inclusion, promote recurrent therapeutic interventions in Portuguese institutions with provide care and supporting services for older adults with dementia, and strengthen research on non-pharmacological therapies. Thus, this multicentre, randomised controlled study is essential to analyse the effects of the individual CS on global cognitive function and specific cognitive domains (e.g., executive functioning, memory) in older adults with mild or moderate AD.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or over.
* Receive care and support services for older adults for at least three months.
* Alzheimer's disease, according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders, 5th edition.
* Ability to communicate and understand.
* Native speakers of Portuguese.
* To have given informed consent for the project, duly completed and signed, after previous information.
* Total scores between 10 and 24 points on the Mini Mental State Examination.

Exclusion Criteria:

* Cannot read and write.
* Severe sensory and physical limitations and/or an acute or serious illness preventing participation in the CS sessions.
* Evidence of aggressive and disruptive behaviour, as indicated by the reference technicians of the institution to which the participant is linked.
* Consumption of psychoactive substances, taking neuroleptics and/or antipsychotics in the last two months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 142 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Cognitive functioning assessed through Mini-Mental State Examination (MMSE) | baseline
  Cognitive functioning assessed by the Mini-Mental State Examination (MMSE), a gold standard screening tool for assessing global cognitive function. Scores range from 0 to 30, with higher scores indicating better cognitive functioning.
Change in cognitive functioning assessed through Mini-Mental State Examination (MMSE) | 12 weeks after the beginning of the intervention
  Change in cognitive functioning evaluated by the Mini-Mental State Examination (MMSE), a gold standard screening tool for assessing global cognitive function.
  Scores range from 0 to 30, with higher scores indicating better cognitive functioning.
Change in cognitive functioning assessed through Mini-Mental State Examination (MMSE) | 12 weeks after end of intervention
  Change in cognitive functioning evaluated by the Mini-Mental State Examination (MMSE), a gold standard screening tool for assessing global cognitive function.
  Scores range from 0 to 30, with higher scores indicating better cognitive functioning.
Cognitive functioning assessed through Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-COG) | baseline
  Evaluates the severity of cognitive deficits in AD in the following domains: memory, orientation, language, praxis and constructive capacity. The total score in the Portuguese version of ADAS-Cog is composed of 11 subtests in the cognitive part and varies between 0 (better performance) and 68 points (worse performance), i.e., higher scores equals better performance.
Change in cognitive functioning assessed through Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-COG) | 12 weeks after the beginning of the intervention
  Evaluates the severity of cognitive deficits in AD in the following domains: memory, orientation, language, praxis and constructive capacity. The total score in the Portuguese version of ADAS-Cog is composed of 11 subtests in the cognitive part and varies between 0 (better performance) and 68 points (worse performance), i.e., higher scores equals better performance.
Change in cognitive functioning assessed through Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-COG) | 12 weeks after end of intervention
  Evaluates the severity of cognitive deficits in AD in the following domains: memory, orientation, language, praxis and constructive capacity. The total score in the Portuguese version of ADAS-Cog is composed of 11 subtests in the cognitive part and varies between 0 (better performance) and 68 points (worse performance), i.e., higher scores equals better performance.
Memory function evaluated through Memory Alteration Test (MAT) | baseline
  The MAT is used to assess memory function. It is an easy and quick instrument that assesses five memory domains: temporal orientation, encoding, semantic memory, free recall, and cued recall. Total scores range from 0 to 50, with higher scores indicating better memory. It has good psychometric properties and is highly sensitive to mild cognitive decline.
Change in memory function evaluated through Memory Alteration Test (MAT) | 12 weeks after the beginning of the intervention
  The MAT is used to assess memory function. It is an easy and quick instrument that assesses five memory domains: temporal orientation, encoding, semantic memory, free recall, and cued recall. Total scores range from 0 to 50, with higher scores indicating better memory. It has good psychometric properties and is highly sensitive to mild cognitive decline.
Change in memory function evaluated through Memory Alteration Test (MAT) | 12 weeks after end of intervention
  The MAT is used to assess memory function. It is an easy and quick instrument that assesses five memory domains: temporal orientation, encoding, semantic memory, free recall, and cued recall. Total scores range from 0 to 50, with higher scores indicating better memory. It has good psychometric properties and is highly sensitive to mild cognitive decline.
Memory function evaluated through Free and Cued Selective Reminding Test (FCSRT) | baseline
  FCSRT is a verbal learning and memory test that allows prompting the encoding and retrieval conditions by using semantic cues on learning and recall trials. It is composed of 16 semantically categorised, unrelated items/words.
Change in memory function evaluated through Free and Cued Selective Reminding Test (FCSRT) | 12 weeks after the beginning of the intervention
  FCSRT is a verbal learning and memory test that allows prompting the encoding and retrieval conditions by using semantic cues on learning and recall trials. It is composed of 16 semantically categorised, unrelated items/words.
Change in memory function evaluated through Free and Cued Selective Reminding Test (FCSRT) | 12 weeks after end of intervention
  FCSRT is a verbal learning and memory test that allows prompting the encoding and retrieval conditions by using semantic cues on learning and recall trials. It is composed of 16 semantically categorised, unrelated items/words.
Executive functions assessed through Frontal Assessment Battery (FAB) | baseline
  FAB assesses executive functions such as abstract thinking, mental flexibility, motor programming, interference sensibility, inhibitory control and environmental independence. Scores range between 0 - 18 points with higher scores indicating better cognitive function.
Change in executive functions assessed through Frontal Assessment Battery (FAB) | 12 weeks after the beginning of the intervention
  FAB assesses executive functions such as abstract thinking, mental flexibility, motor programming, interference sensibility, inhibitory control and environmental independence. Scores range between 0 - 18 points with higher scores indicating better cognitive function.
Change in executive functions assessed through Frontal Assessment Battery (FAB) | 12 weeks after end of intervention
  FAB assesses executive functions such as abstract thinking, mental flexibility, motor programming, interference sensibility, inhibitory control and environmental independence. Scores range between 0 - 18 points with higher scores indicating better cognitive function.
Executive functions assessed through Trail Making Test (TMT) | baseline
  TMT is one of the most widely used instruments in clinical and experimental neuropsychology. It is very sensitive to identify cognitive impairments, measuring simple motor and spatial skills, basic sequencing skills, mental flexibility, selective attention, visuo-perceptual skills, motor speed, and executive functions. Higher scores indicate greater impairment.
Change in executive functions assessed through Trail Making Test (TMT) | 12 weeks after the beginning of the intervention
  TMT is one of the most widely used instruments in clinical and experimental neuropsychology. It is very sensitive to identify cognitive impairments, measuring simple motor and spatial skills, basic sequencing skills, mental flexibility, selective attention, visuo-perceptual skills, motor speed, and executive functions. Higher scores indicate greater impairment.
Change in executive functions assessed through Trail Making Test (TMT) | 12 weeks after end of intervention
  TMT is one of the most widely used instruments in clinical and experimental neuropsychology. It is very sensitive to identify cognitive impairments, measuring simple motor and spatial skills, basic sequencing skills, mental flexibility, selective attention, visuo-perceptual skills, motor speed, and executive functions. Higher scores indicate greater impairment.

OTHER OUTCOMES:
Sociodemographic information gathered through the sociodemographic questionnaire | baseline
  The sociodemographic questionnaire was designed specifically for this study. It gathers information about the participants' gender, age, marital status, educational level, care and support services that the participant attends, medical comorbidities (including cognitive ones), and pharmacological treatment. It will be administered to all participants.
Adherence to the intervention and dropouts evaluated through a session form | during the intervention
  Adherence to the intervention and dropouts will be assessed using a session form, designed specifically for this study, completed by the technician after each session, tracking the attendance and mood/behaviour of the participants throughout the intervention sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Susana I Justo Henriques, PhD, Principal Investigator — Nursing School of Coimbra; Óscar Ribeiro, PhD, Study Director — Aveiro University
Locations (14):
- Portugal (14):
  - Rsocialform - Geriatria, Lda, Mealhada, Aveiro District
  - Santa Casa da Misericórdia da Horta, Açores
  - Cediara - Associação de Solidariedade Social de Ribeira de Fráguas, Aveiro
  - Centro Social e Cultural S. Pedro de Bairro, Braga
  - Centro Social Vale do Homem - Casa da Alegria, Braga
  - Santa Casa da Misericórdia de Castro Marim, Faro
  - Fundação João Bento Raimundo, Guarda
  - Santa Casa da Misericórdia de Alcobaça, Leiria
  - Associação de Socorros da Freguesia de Turcifal, Lisbon
  - Centro de Apoio Social de Oeiras - IASFA, Lisbon
  - Inválidos do Comércio, Lisbon
  - Associação de Apoio Social de Perafita, Porto
  - Santa Casa da Misericórdia de Coruche, Santarém
  - Santa Casa da Misericórdia de Ponte de Lima, Viana do Castelo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Justo-Henriques SI, Silva RCG, Carvalho JO, Perez-Saez E, de Sao Joao RMV, Ribeiro O. Differential response to cognitive stimulation in moderate versus moderately severe Alzheimer's disease. Can J Exp Psychol. 2026 Feb 5. doi: 10.1037/cep0000395. Online ahead of print. PMID 41642798
- [Derived] Justo-Henriques SI, Lemos R, Rahmatpour P, Silva RCG, Carvalho JO, Ribeiro O. Effectiveness of Individual Cognitive Stimulation on Cognition in Mild Alzheimer's Disease: A Multicenter RCT. Psychogeriatrics. 2025 Nov;25(6):e70109. doi: 10.1111/psyg.70109. PMID 41139428